CLINICAL TRIAL: NCT06490939
Title: An Open-label, Parallel-group, Single-center, Phase I Study to Compare the Pharmacokinetic/Pharmacodynamic Characteristics, Safety, and Tolerability of a Single Intravenous Administration of Efepoetin Alfa in Healthy Caucasian and Asian Volunteers
Brief Title: Clinical Trial of Efepoetin Alfa in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GX-E4-HV-003
Record Dates: First submitted 2024-07-01; First posted 2024-07-08 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Asian (Experimental): Single-dose
  Interventions: Drug: Efepoetin Alfa
- Caucasian (Experimental): Single-dose
  Interventions: Drug: Efepoetin Alfa

INTERVENTIONS:
Drug: Efepoetin Alfa — Single-intravenous administration
  Other Names: GX-E4

SUMMARY:
An open-label, parallel-group, single-center, Phase I study to compare the pharmacokinetic/pharmacodynamic characteristics, safety, and tolerability of a single intravenous administration of Efepoetin Alfa in healthy subjects

DETAILED DESCRIPTION:
This study is to objectively evaluate pharmacokinetics as well as pharmacodynamic responses after a single intravenous administration of the Efepoetin alfa, GX-E4, in healthy Caucasian and Asian volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult males and females between the ages of 19-45
2. Asian or Caucasian
3. Body weight >50 kg and <90 kg, BMI 18 ~30 (BMI(kg/m2) = Weight(kg) / {Height(m)}2)
4. Normal hemoglobin range.
5. Normal Serum ferritin and transferrin saturation range.
6. Normal serum folate range
7. Normal vitamin B12 range
8. White blood cell >=3.0 X 10^3 /mm3
9. Platelet >= 150 X 10^3/mm^3 and <450 X 10^3/mm^3
10. Nonsmoker or smoker who smokes below 10 cigarettes a day.

Key Exclusion Criteria:

1. An allergy history, including drug allergies(example: aspirin, antibiotics, etc.) or clinically significant allergy.
2. Liver(including viral hepatitis), renal, respiratory, endocrine, neurological, immunological, blood, psychological, or circulatory system abnormalities, or a history of cancer.
3. Subject who had received EPO, darbepoetin, other EPO supply protein, or immunoglobulin administration, or had received intravenous iron administration.
4. Hypersensitivity to EPO and/or to the excipients of the IMP, or known hypersensitivity to supplementary iron products.
5. Hemoglobinopathy (homozygous sickle cell disease, all types of thalassemia)
6. Systolic blood pressure below 90mmHg or above 140mmHg, or diastolic blood pressure below 50mmHg or above 90mmHg after taking a rest over 3 minutes; pulse rate over 100bpm
7. C-reactive protein level >4mg/dL at 2 weeks prior to the IMP administration.
8. A drug abuse history, or positive in a urine drug-screening test(cocaine, amphetamines, barbiturates, opiates, benzodiazepine, and cannabinoids)
9. Signs of fever, with a temperature of over 38°C, within 1 week before particiation
10. History of epileptic seizure within 6 months before participation
11. Positive to HIV antibody, HBsAg, and HCV antibody test.
12. Consumes over 21 units of alcohol per week, or a person who cannot stay sober for the duration of the entire trial period.
13. Blood donation or a bleeding episode of more than 400mL within 8 weeks prior to study participation
14. The maximum length of the spleen >16cm.
15. Person thought inappropriate by the investigator in consideration of the laboratory test results.
16. Pregnant or breast-feeding.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
PharmacoKinetic parameters (Cmax) | up to 4 weeks
  To measure the concentration of Efepoetin alfa in serum for 336 hours after administration of the investigational product for the pharmacokinetic parameters peak blood concentration
PharmacoKinetic parameters (AUClast) | up to 4 weeks
  To measure the concentration of Efepoetin alfa in serum for 336 hours after administration of the investigational product for the pharmacokinetic parameters area under the blood concentration-time curve

SECONDARY OUTCOMES:
PharmacoKinetic parameters (AUC0-t, AUCinf, AUC%Extrap, CL, tmax, Vd, t1/2) | up to 4 weeks
  Pharmacokinetic parameters of Efepoetin alfa blood concentration after a single intravenous administration of the investigational product
Pharmacodynamic parameters (Emax, ΔEmax, AUEC, ΔAUEC) | up to 4 weeks
  Pharmacodynamic parameters of hemoglobin, reticulocyte and reticulocyte hemoglobin content after administration of the investigational product

OTHER OUTCOMES:
Exploratory | up to 4 weeks
  Assessment or iron storage function
Incidence, nature and severity of adverse events | up to 4 weeks
  Graded according to NCI CTCAE v5.0
Immunogenicity | up to 4 weeks
  Incidence of anti-drug antibodies (ADAs) relative to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No